CLINICAL TRIAL: NCT01986270
Title: A Multicenter, Double-blind, Placebo Controlled, Parallel Group, Study of Two Dose Levels of Oral Eletriptan and Two Dose Levels of of Oral Sumatriptan Given for the Acute Treatment of Migraine
Brief Title: Comparative Study of Oral Eletriptan (40mg and 80mg), Oral Sumatriptan (25mg and 50mg) and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A160-104
Record Dates: First submitted 2013-10-30; First posted 2013-11-18 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Migraine With or Without Aura
MeSH Terms: interventions — eletriptan; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Eletriptan 40 mg (Experimental)
  Interventions: Drug: Eletriptan 40 mg
- Eletriptan 80 mg (Experimental)
  Interventions: Drug: Eletriptan 80 mg
- Sumatriptan 25 mg (Experimental)
  Interventions: Drug: Sumatriptan 25 mg
- Sumatriptan 50 mg (Experimental)
  Interventions: Drug: Sumatriptan 50 mg

INTERVENTIONS:
Drug: Placebo — Matching Placebo
  Arms: Placebo
Drug: Eletriptan 40 mg — 40mg oral
  Arms: Eletriptan 40 mg
Drug: Eletriptan 80 mg — 80mg oral
  Arms: Eletriptan 80 mg
Drug: Sumatriptan 25 mg — 25mg oral
  Arms: Sumatriptan 25 mg
Drug: Sumatriptan 50 mg — 50mg oral
  Arms: Sumatriptan 50 mg

SUMMARY:
The objective of this study was to compare the efficacy, toleration and safety of eletriptan 40mg and 80mg, with sumatriptan 25mg and 50mg, and placebo when given orally to subjects with an acute migraine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who expected to suffer at least one acute attack of migraine, with or without aura, each 6 weeks (The diagnosis of migraine was to comply with the criteria proposed by the International Headache Society (IHS))
* Subjects capable of taking medication as outpatients, and recording the effects of such medication.

Exclusion Criteria:

* Pregnant or breast-feeding women
* Migraine subjects who also suffered from concomitant frequent (non-migrainous) headache, defined as more than six attacks per month on average.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1141 (Actual)
Dates: Start 1996-12; Primary Completion 1998-01 (Actual); Study Completion 1998-01 (Actual)

PRIMARY OUTCOMES:
Headache response at 1 hour after the first dose for the first attack. | 1 hour
  Headache response was defined as improvement from a severe or moderate headache at baseline to either a mild or absent headache post-dose.

SECONDARY OUTCOMES:
Pain-free response at 1 hour after the first dose for the first attack. | 1 hour
  A pain free response was defined as an improvement from a severe or moderate headache at baseline to an absent headache post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A160-104&StudyName=Comparative%20Study%20of%20Oral%20Eletriptan%20%2840mg%20and%2080mg%29%2C%20Oral%20Sumatriptan%20%2825mg%20and%2050mg%29%20and%20Placebo